CLINICAL TRIAL: NCT06196996
Title: Allogeneic Regenerative Islet Transplantation for the Treatment of Brittle Type 1 Diabetes Mellitus: A Clinical Study Evaluating Safety and Efficacy
Brief Title: Allogeneic Regenerative Islet Transplantation for the Treatment of Brittle Type 1 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZXHZ-IIT-02
Record Dates: First submitted 2023-12-13; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Brittle Type 1 Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic Regenerative Islet Transplantation for the Treatment of Brittle Type 1 Diabetes Mellitus (Experimental)
  Interventions: Procedure: The method of islet transplantation is through percutaneous transhepatic portal vein puncture.

INTERVENTIONS:
Procedure: The method of islet transplantation is through percutaneous transhepatic portal vein puncture. — The method of islet transplantation is through percutaneous transhepatic portal vein puncture.After transplantation, rabbit anti human thymocyte immunoglobulin (ATG) or basiliximab was used as induction therapy and low-dose tacrolimus combined with sirolimus or mycophenolate mofetil were used as immunosuppressive maintenance therapy.

SUMMARY:
This is a single-center, single-arm Phase Investigational Intervention Trial (IIT) clinical trial aimed at evaluating the safety and efficacy of allogeneic regenerative islet transplantation for the treatment of brittle type 1 diabetes mellitus. Eighteen patients with brittle type 1 diabetes mellitus, who have inadequate blood glucose control despite intensified exogenous insulin therapy, will be enrolled. The primary endpoint is defined as the safety and improvement in blood glucose levels of the 12 months after allogeneic regenerative islet transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-65 years, gender not specified.
2. Despite intensified exogenous insulin therapy, blood glucose control remains inadequate [glycated hemoglobin ≥7.5%, or TIR (time in range) <70%].
3. Able and willing to use the blood glucose meter provided by the sponsor, conduct self-blood glucose monitoring as required, and complete the patient log as instructed.
4. Fertile eligible subjects (male or female) must agree to use a reliable contraceptive method (hormonal or barrier method or abstinence) during the trial and for at least 90 days after the last dose; premenopausal female patients must have a negative pregnancy test before enrollment.
5. Diagnosed with type 1 diabetes for at least 1 year based on the World Health Organization (WHO) disease diagnostic criteria, and at least one positive result for diabetes-related autoantibodies [glutamic acid decarboxylase autoantibody (GADA), insulinoma-associated-2 autoantibody (IA-2A), insulin autoantibody (IAA), islet cell antibody (ICA), zinc transporter 8 antibody (ZaT8A)]. Experiencing two or more severe hypoglycemic events in the past year, with at least one severe hypoglycemic event in the past 3 months (severe hypoglycemia defined as blood glucose below 2.9 mmol/L or inability to self-correct during hypoglycemia).
6. Voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. Uncontrolled systemic infections, including but not limited to pulmonary tuberculosis, active hepatitis, a history of positive human immunodeficiency virus (HIV) testing, and positive syphilis treponemal antibody (TP);
2. Presence of significant organic lesions in vital organs such as the heart, lungs, or brain;
3. Complications of severe diabetes, including but not limited to retinal hemorrhage, diabetic foot, etc.;
4. Liver function tests with total bilirubin, ALT, and AST ≥2×ULN, and failure to normalize after drug treatment;
5. Untreated cancer or less than 1 year since cure;
6. Severe gastrointestinal dysfunction, gastrointestinal immune diseases, and inability to take immunosuppressant;
7. History of smoking, alcohol abuse, or drug misuse;
8. Severe mental or psychological disorders;
9. Various advanced metabolic diseases (such as hyperuricemia, etc.);
10. Participation in other clinical trials in the 3 months prior to enrollment;
11. Patients requiring long-term oral/intravenous administration of high-dose glucocorticoids due to various diseases;
12. Pregnant or lactating women;
13. Investigator judgment indicating clear evidence of severe, active, uncontrolled endocrine or autoimmune abnormalities other than type 1 diabetes;
14. Other situations judged by the investigator as unsuitable for participation in the trial.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Time in Range | up to 12 months
  Changes in patient blood glucose time in range from baseline
HbA1c | up to 12 months
  Changes in patient HbA1c levels from baseline during the study period
C-peptide | up to 12 months
  Changes in patient fasting and postprandial C-peptide/insulin from baseline during the study period
insulin | up to 12 months
  Changes in patient fasting and postprandial insulin from baseline during the study period

SECONDARY OUTCOMES:
Dose of exogenous insulin | up to 12 months
  Changes in daily exogenous insulin requirements during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yin, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China